CLINICAL TRIAL: NCT00250913
Title: Efficacy and Cost-Effectiveness of Behavioral Counseling For Exercise Behavior in Men and Women Following AMI and PCI
Brief Title: The Efficacy and Cost-Effectiveness of Behavioral Counseling for Exercise in Men and Women Following Acute Myocardial Infarction (AMI) and Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Dr. Robert Reid, Univeristy of Ottawa Heart Insitute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NA 5626
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Arteriosclerosis; Myocardial Infarction
Keywords: motor activity; determinants; psychology; health care costs; quality of life; Angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Motor Activity

INTERVENTIONS:
Behavioral: Telephone-based physical activity counseling program

SUMMARY:
Purpose: The purpose of this project is to determine how effective the telephone-based counseling program is at helping patients with heart disease become more physically active.

Hypotheses to be tested:

* Compared to usual care, patients in the physical activity counseling program will:

  1. significantly increase total distance measured by an accelerometer and minutes of physical activity at a moderate intensity or higher,
  2. have significantly higher generic and heart-disease health-related quality of life, and
  3. will lead to greater improvements in the mediators of behavior change (psychosocial variables, i.e. self-efficacy, outcome expectations, etc.) at 26 and 52 weeks;
* Changes in the mediators of physical activity will predict changes in physical activity outcomes at 26 and 52 weeks;
* The physical activity counseling program is preferable to usual care from the perspective of health care system costs.

DETAILED DESCRIPTION:
Most existing cardiac rehabilitation programs have little ability to expand participation using traditional delivery models that emphasize supervised, facility-based programs. Furthermore, facility-based programs to promote physical activity behavior in patients with coronary artery disease (CAD) are limited in their impact because most patients are unwilling to travel more than 30-45 minutes to participate in a program. The University of Ottawa Heart Institute Prevention and Rehabilitation Centre (Ottawa, Canada) has developed a telephone-based counseling program, specifically to support heart patients in becoming more physically active. The study will involve patients either participating in a 12-month physical activity counseling (PAC) program, or receiving usual care after they are discharged from hospital. For patients assigned to the PAC group, a face-to-face meeting with a physical activity counselor will occur within 10 days to 2 weeks after being discharged from hospital. At this time the patient will be provided with a personalized physical activity program which will be tailored based on prior activity levels, clinical history, and recovery. The PAC patients will also receive eight telephone-based counseling sessions at 2, 4, 8, 14, 20 and 24 weeks, and 2 telephone maintenance contacts at 40 and 52 weeks after hospital discharge. Each telephone call is scheduled to last 10-15 minutes. For patients assigned to the usual care (UC) group, they will receive the physical activity advice and care usually provided to patients discharged from hospital. Following hospitalization, usual care typically includes a follow-up visit(s) with your cardiologist and/or family doctor. If requested, an activity program will be provided to usual care group participants after the study has finished. In addition, the patients will also be required to complete five research questionnaires, and two telephone interviews. The study will track all participants for a period of one year from the time they are discharged from hospital. Over the next twelve months 252 patients from the Ottawa Heart Institute are expected to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Diagnosis:

  1) hospitalized patients ready for discharge following successful PCI procedure
* Including patients receiving PCI following admission for AMI or hospitalized post-AMI patients who have not been revascularized
* No lesions with >50 % stenosis
* English proficiency in reading, writing and speaking
* Age: 20-85 years

Exclusion Criteria:

* Those patients who are already taking part in another research trial.
* Patient intends to enroll, or is currently enrolled in structured cardiac rehabilitation
* Unable to participate in the on-site cardiac supervised rehab program, cardiac rehab lite, case-managed home cardiac rehab program, Pembroke cardiac rehab program
* Hospitalization for coronary artery bypass (CABG)
* Chronic obstructive pulmonary disease (COPD)
* Hospitalization for diagnostic procedure not associated with previously documented MI
* Patient coming back to hospital for planned staged PCI within 6 months
* Cardiac transplantation
* Presence of, or hospitalization for defibrillator implant
* Hospitalization for pacemaker implantation
* Unresolved unstable angina and/or hospitalization for angina (without MI or PCI)
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Neuromuscular, musculoskeletal or rheumatoid disorders that are exacerbated by exercise
* Other uncontrolled metabolic conditions (e.g. diabetes)
* Chronic infectious diseases such as mononucleosis, hepatitis, AIDS
* Acute systemic illness or fever
* Uncontrolled tachycardia (<120 bpm)
* Uncompensated congestive heart failure (and/or NYHA Class III, or IV)
* 3rd degree atrioventricular (AV) block (without pacemaker)
* Active pericarditis or myocarditis
* Recent embolism
* Suspected or known abdominal aortic aneurysm (AAA) > 4cm
* Uncontrolled hypertension (systolic blood pressure [SBP] >200; diastolic blood pressure [DBP] >110)
* Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
7-day physical activity levels: waist mounted pedometer will be worn to measure distance (km) over a period of 9 days and will be recorded in an activity log, as well as, reported intensity and duration of activities at a moderate level+
7-day physical activity recall (PAR): interview administered following the pedometer wear to verify the completeness of the patient recorded activity log and to account for leisure and occupational/domestic activities
Primary outcomes measured at baseline and 6 and 12 months

SECONDARY OUTCOMES:
Psychosocial and Environmental Mediators (questionnaire): psychosocial and environmental mediators of physical activity
Quality of Life (questionnaire): heart disease health-related quality of life
generic quality of life
secondary outcomes measured at baseline and 6 and 12 months
Health Care Systems Costs (questionnaire and telephone): the costs of in-person and telephone-based behavioral counseling sessions and any additional health care relating to coronary artery disease (CAD)
the use of health care resources will be measured for medical event updates, patient related costs and work absenteeism
cost utility analysis to assess for cost per quality-adjusted life year (QALY)
measured at 3 (telephone), 6 (questionnaire), 9 (telephone) and 12 (questionnaire) months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, PhD, MBA, Principal Investigator — Ottawa Heart Institute Research Corporation; Louise Morrin, RPT, MBA, Study Chair — Ottawa Heart Institute Research Corporation; Lyall Higginson, MD, FRCP(C), Study Chair — Ottawa Heart Institute Research Corporation; Andrew Pipe, MD, Study Chair — The University of Ottawa Heart Institute; Andreas Wielgosz, MD, FRCP(C), Study Chair — The Ottawa General Hospital - Department of Cadiology - General Campus; Neil Oldridge, PhD, Study Chair — College of Health Sciences, University of Wisconsin-Milwaukee; George Wells, PhD, Study Chair — Clinical Epidemiology Unit, University of Ottawa Heart Institute; Chris Blanchard, PhD, Study Chair — Department of Human Kinetics, University of Ottawa & University of Ottawa Heart Institute
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Baranowski T, Anderson C, Carmack C. Mediating variable framework in physical activity interventions. How are we doing? How might we do better? Am J Prev Med. 1998 Nov;15(4):266-97. doi: 10.1016/s0749-3797(98)00080-4. PMID 9838973
- [Background] Arthur HM, Smith KM, Kodis J, McKelvie R. A controlled trial of hospital versus home-based exercise in cardiac patients. Med Sci Sports Exerc. 2002 Oct;34(10):1544-50. doi: 10.1097/00005768-200210000-00003. PMID 12370553
- [Background] Drummond M, O'Brien BJ, Stoddart G, Torrance G. Methodsfor the Economic Evaluation of Health Care Programmes:Oxford Medical Publications; 1997.
- [Background] Thompson PD, Buchner D, Pina IL, Balady GJ, Williams MA, Marcus BH, Berra K, Blair SN, Costa F, Franklin B, Fletcher GF, Gordon NF, Pate RR, Rodriguez BL, Yancey AK, Wenger NK; American Heart Association Council on Clinical Cardiology Subcommittee on Exercise, Rehabilitation, and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism Subcommittee on Physical Activity. Exercise and physical activity in the prevention and treatment of atherosclerotic cardiovascular disease: a statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity). Circulation. 2003 Jun 24;107(24):3109-16. doi: 10.1161/01.CIR.0000075572.40158.77. No abstract available. PMID 12821592
- [Background] Centres for Disease Control. Physical activity and health: Areport of the Surgeon General. Atlanta: National Centre forChronic Disease Prevention and Health Promotion; 1999.
- [Background] Stone JA, Cyr C, Friesen M, Kennedy-Symonds H, Stene R, Smilovitch M; Canadian Association of Cardiac Rehabilitation. Canadian guidelines for cardiac rehabilitation and atherosclerotic heart disease prevention: a summary. Can J Cardiol. 2001 Jun;17 Suppl B:3B-30B. PMID 11420586
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Sallis JF, Johnson MF, Calfas KJ, Caparosa S, Nichols JF. Assessing perceived physical environmental variables that may influence physical activity. Res Q Exerc Sport. 1997 Dec;68(4):345-51. doi: 10.1080/02701367.1997.10608015. PMID 9421846
- [Background] King AC, Stokols D, Talen E, Brassington GS, Killingsworth R. Theoretical approaches to the promotion of physical activity: forging a transdisciplinary paradigm. Am J Prev Med. 2002 Aug;23(2 Suppl):15-25. doi: 10.1016/s0749-3797(02)00470-1. PMID 12133734